CLINICAL TRIAL: NCT02191358
Title: YouScript IMPACT (Improving Medication Protocols and Abating Cost of Treatment) Registry
Brief Title: YouScript IMPACT Registry
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Genelex Corporation (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: Genelex 2014-01
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2015-09

CONDITIONS: Adverse Drug Events; Adverse Drug Reactions; Drug Interaction Potentiation; Drug Metabolism, Poor, CYP2D6-RELATED; Drug Metabolism, Poor, CYP2C19-RELATED; Cytochrome P450 Enzyme Deficiency; Cytochrome P450 CYP2D6 Enzyme Deficiency; Cytochrome P450 CYP2C9 Enzyme Deficiency; Cytochrome P450 CYP2C19 Enzyme Deficiency; Cytochrome P450 CYP3A Enzyme Deficiency; Poor Metabolizer Due to Cytochrome P450 CYP2C9 Variant; Poor Metabolizer Due to Cytochrome P450 CYP2C19 Variant; Poor Metabolizer Due to Cytochrome P450 CYP2D6 Variant
Keywords: Cytochrome drug interactions; Drug-drug interaction; Drug-gene interaction; Drug-drug-gene interaction; Drug Metabolism; Elderly; Geriatric medicine; Geriatrics; Personalized medicine; Pharmacist; Pharmacogenetics; Pharmacogenomics; Pharmacokinetics; Polymorphism; Polypharmacy; Precision medicine; Seniors; YouScript; CYP2C9; CYP2C19; CYP2D6; CYP3A4; CYP3A5; VKORC1; Amitriptyline; Aripiprazole; Atomoxetine; Carvedilol; Celecoxib; Citalopram; Clobazam; Clomipramine; Clopidogrel; Clozapine; Codeine; Desipramine; Dextromethorphan; Diazepam; Doxepin; Escitalopram; Esomeprazole; Fesoterodine; Flecainide; Fluoxetine; Flurbiprofen; Fluvoxamine; Haloperidol; Hydrocodone; Ibuprofen; Iloperidone; Imipramine; Indomethacin; Meloxicam; Metoprolol; Mexiletine; Nortriptyline; Omeprazole; Oxycodone; Paroxetine; Perphenazine; Phenobarbital; Phenytoin; Pimozide; Piroxicam; Proguanil; Propafenone; Propranolol; Risperidone; Sertraline; Tetrabenazine; Thioridazine; Timolol; Tolterodine; Torsemide; Tramadol; Trimipramine; Venlafaxine; Voriconazole; Vortioxetine
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Drug Metabolism, Poor, CYP2D6-Related; Drug Metabolism, Poor, CYP2C19-Related; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- "Tested" patients (prospective): Patients whose providers decide to have them undergo testing via the YouScript Personalized Prescribing System will be recruited for the study. Data will be gathered at baseline and 120 days later. The decision to utilize YouScript and all treatment decisions will be made at the discretion of the provider in accordance with their usual care practice, and will be made prior to the decision to participate in the study.
- "Untested" patients (retrospective): Patients for comparison to the prospectively followed patients will be derived from Inovalon's MORE2 healthcare database. Patients meeting the same enrollment criteria (excluding the YouScript testing) will be matched on key characteristics to the tested patients. Outcomes will be compared between the prospectively enrolled patients undergoing pharmacogenetic testing with the YouScript Personalized Prescribing System at the discretion of their treating physician.

SUMMARY:
This multicenter observational study aims to investigate the benefits of providing pharmacogenetic testing with the YouScript Personalized Prescribing System which includes a clinical decision support tool and individualized pharmacist recommendations to elderly polypharmacy patients who are most at risk of adverse drug events. The YouScript system is unique in identifying drug-gene, and drug-drug-gene interactions that are missed by existing systems, and represent over 35% of significant interaction warnings. Data analysis will assess the impact of recommendations for medication changes on clinical decision making, patient outcomes, and healthcare resource utilization to determine which medications, specialties, or patient segments derive the greatest benefit from this intervention. Data gathered from patients enrolled in this study will be compared to patients matched on key characteristics from Inovalon's MORE2 healthcare database.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Genelex Corporation is a leader in comprehensive medication management based on the YouScript clinical decision support tool and DNA drug sensitivity testing. Controlling prescription drug adverse event risk is complex because more than 85% of patients have significant DNA based variation in activity of the cytochrome p450 (CYP) enzymes that metabolize the majority of the most commonly prescribed medicines. Polypharmacy, common in the elderly and chronically ill further increases the risk of an adverse drug event (ADE). The public healthcare problem resulting from these factors costs an estimated $289 billion per year in excess health care costs.

The goal of the YouScript personalized prescribing system is to improve patient outcomes by preventing ADEs caused by drug-drug, drug-gene and drug-drug-gene interactions. ADEs are defined to include prescription and over-the-counter (OTC) drug overdose toxicity, adverse drug reactions (ADRs), and treatment failures generally caused by properly prescribed medications. The YouScript system prevents ADEs by the combined analysis of patient drug regimens and individual genetics. YouScript DNA drug sensitivity testing includes five enzymes in the cytochrome P450 (CYP) group (CYP2D6, CYP2C9, CYP2C19, CYP3A4, and CYP3A5). YouScript synthesizes decades of publicly funded basic and clinical research to provide actionable information to physicians treating patients.

Elderly patients are at greater risk of an ADE. Two-thirds of adults age 65 or older take one or more prescription drugs daily. Patients age 60 years and older account for 10-17% of hospitalizations and 51% of the deaths from ADEs, although this age group represents just 17% of the U.S. population. Following discharge, 50% of patients with ADRs declined in one or more activities of daily living, compared to 24% of patients without ADRs.

Although the value of pharmacogenetic testing and comprehensive gene-based medication management is being recognized by clinicians, it is still not endorsed by many expert committees and third party payers for most prescription drugs. The purpose of this study is to meet the need for evidence that better demonstrates the impact of such comprehensive gene-based medication management on healthcare resource utilization (HRU), clinical decision-making, and patient outcomes. Therefore, the proposed study aims to assess the impact of the YouScript Personal Prescribing System on HRU, clinical decision-making, and clinical outcomes.

OBJECTIVES:

Primary objective:

To determine the impact of the YouScript Personalized Prescribing System on HRU.

Secondary objectives:

To assess the impact of the YouScript Personalized Prescribing System on clinical decision-making, including risk modification through dosage adjustment and medication change.

To assess the impact of the YouScript Personalized Prescribing System on the number of ADEs experienced by patients.

STUDY DESIGN:

The study is designed as a prospective, non-interventional, observational study to assess the real-world impact of the YouScript Personalized Prescribing System on HRU, provider clinical decision-making, and ADEs. The decision to utilize the YouScript Personalized Prescribing System and all treatment decisions will be made in accordance with usual care practice, and will be made prior to the decision to participate in the study.

Outcomes will be compared between a group of prospectively enrolled patients undergoing CYP2D6, CYP2C19, CYP2C9, VKORC1, CYP3A4, and CYP3A5 testing with the YouScript Personalized Prescribing System at the discretion of their provider (i.e. "tested" patients) and data from a group of similar patients included in Inovalon's MORE2 healthcare database meeting the same enrollment criteria (excluding the YouScript testing) and matched on key characteristics to the tested patients using propensity score matching. Sites will be queried regarding use of other drug-drug interaction (DDI) systems to better distinguish the impact of YouScript vs. other systems.

The study aims to initially enroll 1500 patients from 3-15 sites in the United States, identified by Genelex. The study may be expanded up to 10,000 patients at additional sites in the United States. The study duration is estimated to be at least 15 months, including 3 months for study set-up, 6 months or longer for patient enrollment depending on the rate of accrual at each site, 4 months of per-patient follow-up and 2 months for study closeout.

A pilot study consisting of the first 150 patients enrolled will be conducted prior to continuing enrollment in order to assist with planning the larger-scale study, such as confirming appropriate length of follow-up necessary to observe patient outcomes, comparison of patient baseline characteristics, identifying potential variables for propensity score matching, sample size calculation, and necessary changes to case report forms.

After a discussion about the study with study staff and providing informed consent, baseline data will be collected (described in more detail below), including a buccal swab or blood sample, from patients undergoing YouScript testing. Follow-up data will be collected 120 days after enrollment on all patients. Patients will be seen in the clinic or phoned (if a visit is not scheduled in 120 days ± 14 days from baseline) and queried regarding HRU (including number of hospitalizations, ER visits, provider office visits, and procedures), changes in medications, reason for changes, and adverse drug events. This data will also be abstracted from the medical record for completeness. In addition, providers utilizing YouScript will also be surveyed regarding the usefulness of YouScript in their clinical decision-making.

Similar available data will be abstracted for a sample of presumably untested patients included in the MORE2 registry database who meet eligibility criteria and are matched to prospectively enrolled patients on key characteristics using propensity score matching.

CLINICAL ASSESSMENTS:

As this is an observational study, there are no mandatory visits. While the timing of actual patient visits will occur at the discretion of the treating provider, it will be requested that data be entered at baseline and again 120 days after enrollment regardless of the number of times that a patient had been seen during that interval. All data will be collected and entered by the sites directly into a web-based electronic data capture (EDC) system via electronic case report forms (eCRFs).

After patients are screened and consented, the following variables will be collected at baseline, with some being collected as part of the standard YouScript requisition form: demographics, current smoking status, active medical conditions, liver or kidney dysfunction, drugs of interest and other concomitant medications (including date of initiation of therapy, dose, frequency, and indication, respectively), previous ADEs to any drug of interest, and buccal swab/blood sample for YouScript testing. The site will not be required to enter data collected on the YouScript requisition form into the eCRF.

The following follow-up data will be collected during a routinely scheduled visit, or by phone if a visit is not scheduled, approximately 120 days after enrollment: number of hospitalizations; ER visits, diagnostic or surgical procedures, and office visits since baseline; Change/consider/monitor recommendations for drug regimen change(s) by the pharmacy team; changes in drug regimen/dose for drugs of interest and concomitant medications since baseline; reason for changing or not changing drug regimen/dose; ADEs since baseline; and healthcare provider survey/questions regarding role and usefulness of YouScript in clinical decision making. If a visit is not scheduled at 120 days ±14 days, the study staff will contact patients by telephone and data will be collected. If patients choose to terminate participation before completion of the 120-day follow---up, all follow-up data will be collected, as well as the reason for discontinuation.

DATA ANALYSIS:

Complete analytical specifications, including tables and listings, will be fully detailed in the statistical analysis plan (SAP). Descriptive analyses will be performed to gain an understanding of the qualitative and quantitative nature of the data collected and the characteristics of the sample studied. Summary statistics will be calculated and presented for baseline characteristics and outcomes for tested and control groups separately.

Comparative analyses will be conducted to determine whether there are statistically significant differences in specific quantitative outcomes between tested and control groups. Because of propensity score matching between tested and control patients, unadjusted comparative analysis will be performed and reported as the primary results. Adjusted analysis using multiple regression models will be used to examine potential confounding effects that cannot be addressed by the matching process. Exploratory analyses will be conducted to explore the impact of YouScript in various subgroups and to identify potential subgroups which will be most likely to benefit from YouScript, as deemed appropriate.

The first interim analysis will be conducted after data collection is complete for approximately the first 150 prospectively enrolled patients (i.e. the pilot study) to determine if any changes are necessary in the methods of the larger scale study. The second interim analysis will be completed after data collection is complete for approximately 750 prospectively enrolled patients.

For the main analyses, differences in HRU at the 120-day follow-up will be determined by comparing the mean number of hospitalizations, emergency room visits, diagnostic procedures, surgical procedures, and clinic visits between the tested and untested groups. The impact of YouScript on clinical decision making will be determined by comparing the mean number of changes in drug regimen or dose between those who underwent YouScript testing and those that did not. In addition, the number of ADEs experienced by patients during the 120-day study will be compared between the tested and untested groups. Comparisons will be made with the t-test (if the data are normally distributed), the Wilcoxon-Rank-Sum test (if the data are continuous and not normally distributed), or the chi-squared (or Fisher exact) test if the data are considered categorical. Multivariable linear regression models will be used to examine the association of the YouScript Personalized Prescribing System with HRU, clinical decision making, and ADEs, respectively, while controlling for potential confounding effects from baseline characteristics not included in the propensity score matching process.

In tested patients only, HRU, number of ADEs, and number of changes in drug regimen/dose will be examined in relationship to genotype, sample size permitting. Reasons for not changing drug regimen or dose when a recommendation was made will be summarized qualitatively or be analyzed quantitatively if possible. In addition, calculation of the drug-gene, drug-drug-gene and drug-drug interaction recommendation acceptance rate (as defined by whether a drug or dose was changed after a recommendation was made) will be calculated. Provider feedback regarding whether the YouScript Personalized Prescribing System impacted their clinical decisions will be summarized quantitatively and qualitatively.

ELIGIBILITY:
INCLUSION CRITERIA: Prospectively enrolled study participants (i.e. "tested" patients) must fulfill all of the following criteria to be eligible for enrollment into the study:

* Age 65 or older
* Willing and able to provide informed consent for study participation either directly or by a legally authorized representative (LAR)
* Undergoing testing through the YouScript Personalized Prescribing System as recommended during the course of routine care, and ordering all of the following tests: CYP2D6, CYP2C19, CYP2C9, VKORC1, CYP3A4, CYP3A5
* Currently taking at least 3 prescription medications (any route of administration)
* Initiated treatment with, or changed the dose of, at least 1 of the following oral forms of medication (excluding medications taken PRN) within the previous 120 days (generic name given with major U.S. brand name given in parentheses). These medications are subject to significant drug---gene interactions as defined by FDA boxed warning, FDA cautionary labeling, clinical literature or a YouScript algorithm---predicted significant effect:

Amitriptyline (Elavil), Aripiprazole (Abilify), Atomoxetine (Strattera), Carvedilol (Coreg), Celecoxib (Celebrex), Citalopram (Celexa), Clobazam (Onfi), Clomipramine (Anafranil), Clopidogrel (Plavix), Clozapine (Clozaril), Codeine [Tylenol #3 (combo)], Desipramine (Norpramin), Dextromethorphan (Delsym), Diazepam (Valium), Doxepin (Sinequan), Escitalopram (Lexapro), Esomeprazole (Nexium), Fesoterodine (Toviaz), Flecainide (Tambocor), Fluoxetine (Prozac), Flurbiprofen (Ansaid), Fluvoxamine (Luvox), Haloperidol (Haldol), Hydrocodone (Zohydro), Ibuprofen (Motrin), Iloperidone (Fanapt), Imipramine (Tofranil), Indomethacin (Indocin), Meloxicam (Mobic), Metoprolol (Toprol-XL), Mexiletine (Mexitil), Nortriptyline (Pamelor), Omeprazole (Prilosec), Oxycodone (Oxycontin), Paroxetine (Paxil), Perphenazine (Trilafon), Phenobarbital (Luminal), Phenytoin (Dilantin), Pimozide (Orap), Piroxicam (Feldene), Proguanil [(Malarone (combo)], Propafenone (Rythmol), Propranolol (Inderal), Risperidone (Risperdal), Sertraline (Zoloft), Tetrabenazine (Xenazine), Thioridazine (Mellaril), Timolol (Apotimol), Tolterodine (Detrol), Torsemide (Demadex), Tramadol (Ultram), Trimipramine (Surmontil), Venlafaxine (Effexor), Voriconazole (Vfend), Vortioxetine (Brintellix)

For a list of the inclusion criteria adapted to the "untested" patients (retrospective cohort), see the protocol.

EXCLUSION CRITERIA: Patients (prospective and retrospective) meeting any of the following criteria will not be eligible for enrollment/inclusion in the study (ICD9 codes are included for retrospective database patients):

* Previous CYP testing (CPT codes 81225, 81226, 81227)
* History of organ transplant (199.2; 238.77; 414.06; 414.07; 996.80---996.89; E878.0; V42.0---V42.7; V42.81---V42.84; V42.89; V42.9; V45.87; V49.83; V58.44)
* Patient currently receiving intravenous antibiotics
* Currently taking immunosuppressants (azathioprine, cyclosporine, monoclonal antibodies, corticosteroids)
* Current malabsorption syndrome (579.0), including the following: Intestinal malabsorption (579.8, 579.9), Postoperative malabsorption (579.3), Short bowel syndrome (579.3)
* Current hospitalization
* Treatment of invasive solid tumors or hematologic malignancies in the last year, excluding in situ cancers or non-melanoma skin cancer (basal cell carcinoma)
* Currently malnourished, as determined by treating provider

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study consists of patients age 65 and older who are currently on or initiating treatment with at least one oral form of medication (excluding medications taken PRN) with a significant drug-gene interaction as defined by black box warning, FDA cautionary labeling, clinical literature or a YouScript algorithm-predicted significant effect. Those meeting eligibility criteria and undergoing YouScript testing according to their provider's usual care practice will be eligible for prospective enrollment into the "tested" group. Those included in Inovalon's MORE2 healthcare database meeting enrollment criteria between January 1, 2013 and June 30, 2013 will be eligible for inclusion in the "untested" group.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Healthcare Resource Utilization | 120 days
  The primary objective is to determine the impact of the YouScript Personalized Prescribing System on healthcare resource utilization. This will involve comparing the number of hospitalizations, number of ER visits, number of provider office visits, number of radiographic procedures, and number of surgeries for the tested group versus the untested group.

SECONDARY OUTCOMES:
Clinical decision-making | 120 days
  A secondary objective is to assess the impact of the YouScript Personalized Prescribing System on clinical decision-making, including risk modification through dosage adjustment. This will involve comparing changes in drug regimen/dose, as well as reasons for any changes and healthcare provider survey/question regarding the role and usefulness of YouScript in clinical decision making/or medication change for the tested group versus the untested group.
Adverse Drug Events | 120 days
  A secondary objective is to assess the impact of the YouScript Personalized Prescribing System on the number of adverse drug events experienced by patients. This will involve comparing the number of adverse events experienced by patients along with severity and relatedness for the tested group versus the untested group.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Brixner, PhD, RPh, Principal Investigator — University of Utah
Locations (7):
- United States (7):
  - Dr. Michael Dao, Garden Grove, California
  - Kaiser Permanente Colorado, Denver, Colorado
  - Gill Heart Institute, Lexington, Kentucky
  - IRC Clinics, Towson, Maryland
  - Internal Medicine & Cardiology Associates, Fall River, Massachusetts
  - Prima CARE, Fall River, Massachusetts
  - Carilion Clinic, Christiansburg, Virginia

REFERENCES:
- [Result] Brixner D, Biltaji E, Bress A, Unni S, Ye X, Mamiya T, Ashcraft K, Biskupiak J. The effect of pharmacogenetic profiling with a clinical decision support tool on healthcare resource utilization and estimated costs in the elderly exposed to polypharmacy. J Med Econ. 2016;19(3):213-28. doi: 10.3111/13696998.2015.1110160. Epub 2015 Nov 11. PMID 26478982
- See also: Sponsor website — http://genelex.com
- See also: Genelex Publishes Study Hoping to Improve PGx Panel Test Reimbursement; Medicare Remains Unconvinced — https://www.genomeweb.com/molecular-diagnostics/genelex-publishes-study-hoping-improve-pgx-panel-test-reimbursement-medicare